CLINICAL TRIAL: NCT04498884
Title: Double-blinded, Randomized, Comparative, Crossover Study of the Pharmacokinetics of Rinsulin® Mix 30/70, Suspension for Subcutaneous Administration, 100 IU / ml (OJSC GEROPHARM-Bio, Russia) and Humulin® M3, Suspension for Subcutaneous Administration, 100 IU / ml (Lilly France, France) Using the Method of Euglycemic Hyperinsulinemic Clamp on Healthy Volunteers
Brief Title: Comparative Study of the Pharmacokinetics of Rinsulin® Mix 30/70, Suspension for Subcutaneous Administration, 100 IU / ml (OJSC GEROPHARM-Bio, Russia) and Humulin® M3, Suspension for Subcutaneous Administration, 100 IU / ml (Lilly France, France) Using the Euglycemic Hyperinsulinemic Clamp Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RIN30-70-CL
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Bioequivalence
Keywords: human recombinant insulin; euglycemic hyperinsulinemic clamp

STUDY DESIGN:
Intervention Model Description: two-period two-way crossover
Who Masked: Participant, Investigator
Masking Description: douuble-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rinsulin® mix 30/70 (Experimental): Single subcutaneous administration of Insulin at a dose 0.4 IU / kg
  Interventions: Drug: Rinsulin® mix 30/70; Drug: Humulin® M3
- Humulin® M3 (Active Comparator): Single subcutaneous administration of Insulin at a dose 0.4 IU / kg
  Interventions: Drug: Rinsulin® mix 30/70; Drug: Humulin® M3

INTERVENTIONS:
Drug: Rinsulin® mix 30/70 — one subcutaneous injection at a dose of 0.4 IU/kg
Drug: Humulin® M3 — one subcutaneous injection at a dose of 0.4 IU/kg

SUMMARY:
Pharmacokinetics and pharmacodynamics study of 2 formulations of insulin mixtures Rinsulin® Mix 30/70, Suspension for Subcutaneous Administration, 100 IU / ml (OJSC GEROPHARM-Bio, Russia) versus Humulin® M3, Suspension for Subcutaneous Administration, 100 IU / ml (Lilly France, France).

DETAILED DESCRIPTION:
Double-blinded, randomized, comparative, crossover study of comparative pharmacokinetics of Rinsulin® mix 30/70, suspension for subcutaneous administration, 100 IU / ml (OJSC GEROPHARM-Bio, Russia) and Humulin® M3, suspension for subcutaneous administration, 100 IU / ml (Lilly France, France) using hyperinsulinemic euglycemic clamp method on healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent to participate in the study.
* Men of the Caucasian race with a verified diagnosis "healthy" according to the data of standard clinical, laboratory and instrumental examination methods.
* Age 18-50, inclusive.
* Body mass index 18.5 - 27 kg / m2.
* Volunteers who have sexual contact with fertile women should agree to use barrier methods of contraception while participating in the study (unless they have undergone surgical sterilization). Study Participants must also not become a sperm donor within the specified period.
* Consent to all restrictions imposed during the study.

Exclusion Criteria:

* Acute inflammatory diseases within 3 weeks from the moment of complete recovery to the stage of screening.
* Presence in the family history of the closest relatives cases of verified diagnosis of diabetes mellitus of any type.
* Deviations from the norm of basic vital indicators (heart rate, blood pressure, respiratory rate, body temperature) and ECG from normal values and laboratory values from reference values during screening.
* Fasting plasma glucose> 6.1 mmol / L at screening.
* HbA1C> 6% at the time of screening.
* Oral glucose tolerance test - blood glucose level ≥7.8 mmol / L (2 hours after glucose loading) during screening.
* Hard-to-reach veins of the upper extremities, vein thrombosis, history of thrombophlebitis or family history of close relatives, "compromised" veins due to frequent preceding venipuncture.
* Taking medications, phytopreparations, biologically active additives within 14 days before screening.
* Significant blood loss 3 months before screening due to, for example, but not limited to the following points: a. donor blood donation; b. extended surgery or trauma leading to significant blood loss.
* Incomplete recovery from surgery or surgery scheduled while the volunteer is participating in the study.
* Mental, physical and other reasons interferes with adequately assessing behavior and correctly fulfill the conditions of the research protocol incl.:

  1. A history of mental illness;
  2. Current or history (three years before the first administration of the study drug) of narcotic, drug and / or substance abuse. A positive test for the content of drugs in urine during the screening period;
  3. Anamnestic information about alcoholism or intake of more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of dry wine or 50 ml of spirits). A positive test for alcohol in breath during the screening period;
  4. Nicotine addiction (regular use of tobacco less than 6 months before screening).
* Any chronic diseases, incl. but not limited to positive test results for hepatitis C or hepatitis B, HIV, syphilis at the time of screening, Burdened allergological history.
* Presence of suspicion of an inflammatory disease of the urinary system based on the results of urinalysis during screening.
* Presence of oncological diseases within 5 years before the screening.
* History of organ transplantation (except of corneal transplant performed more than 3 months before the first injection of the study drug).
* Participation in a clinical trial of any drug or experimental medical device within 3 months prior to the first administration of the study drug.
* Any other condition that, in the reasonable opinion of the research physician, makes it difficult for the volunteer to participate in the study.
* History of hypersensitivity to heparin, insulin or any of the excipients of the investigational drugs.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
AUC 0-12 | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Total area under the curve "drug concentration - time" in the time interval from 0 to 12 h
Cmax | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Test Drug Observed Maximum Plasma Concentration
GIR 0-12 | 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 12 h
GIR 0-24 | 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Total area under the curve "glucose infusion rate - time" in the time interval from 0 to 24 h
GIR max | 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Maximum glucose infusion rate over the study period
tGIRmax | 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Time to reach maximum glucose infusion rate
TGIRlag | 1, -0.5, then every 5 min till 10 hour, every 10 min till 12 hour, every 15 min till 24 hour
  Time between the drug administration and the onset of action

SECONDARY OUTCOMES:
AUC 0-2 | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Total area under the curve "drug concentration - time" in the time interval from 0 to 2 h
AUC 0-24 | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Total area under the curve "drug concentration - time" in the time interval from 0 to 24 h
AUC 0-6 | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Total area under the curve "drug concentration - time" in the time interval from 0 to 6 h
AUC 0-∞ | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Total area under the curve "drug concentration - time" in the time interval from 0 h to ∞
mean residence time | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  average residence time of a drug molecule in the body
kel | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  constant for drug elimination rate
Tmax | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Time to reach test drug Maximum Plasma Concentration
t1/2 | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  Half-life of a drug tested
t50%-early | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  reaching 50% of the maximum insulin concentration before reaching Cmax
t50%-late | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  reaching 50% of the maximum insulin concentration after reaching Cmax
ratio Сmax/AUC0-t | -0.5 , 0, every 15 min till 6 h, every 30 min till 11h, every 60 min till 17h, every 120 min till 24h
  relative absorption rate

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - "National Medical Research Center of Endocrinology" of the Ministry of Health of the Russian Federation, Moscow
  - National Medical Research Center in name of V.A. Almazov " of the Ministry of Health of the Russian Federation, Saint Petersburg
  - LLC "BioEk", Russian Federation, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No